CLINICAL TRIAL: NCT04300023
Title: Examining the Reach, Effectiveness and Maintenance of Social Engagement on Exercise Outcomes: In-home Cycling for Individuals With Parkinson Disease
Brief Title: In-home Cycling for Individuals With PD: Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0414: Feasibility; A176000 (Other: UW Madison); EDUC\KINESIOLOGY\KINESIO (Other: UW Madison); 1UL1TR002373-01 (NIH); 1KL2TR002374-01 (NIH)
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: social support; exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: 12 participants randomly assigned to social cycling group or solo cycling group, solo group participants crossed over to the social group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solo Cycling Control Group (No Intervention): Exercise bike delivered to their home, custom fit to their needs and installed in a safe location. Participants will be provided with exercise recommendations, but will receive only data recording calls every 2-weeks. [will crossover and complete the cycling intervention following the initial 6-months]
- Social Cycling Group (Experimental): Exercise bike delivered to their home, custom fit to their needs and installed in a safe location, sessions will consist of up to 30 minutes of cycling while engaged in social interaction with a research staff member, thus providing a social/community aspect that would not otherwise be present.
  Interventions: Behavioral: Social Cycling Group

INTERVENTIONS:
Behavioral: Social Cycling Group — engaged with a research staff member for 30 minutes of cycling
  Arms: Social Cycling Group

SUMMARY:
This study will examine the influence of social support on exercise frequency, duration, quality of life, and overall activity level.

DETAILED DESCRIPTION:
The benefits of exercise for individuals with Parkinson disease (PD) have been well documented; however, individuals with PD living in rural and underserved urban settings are largely unable or unwilling to participate in group exercise programs due in large part to their distance from such programs and financial considerations. Additionally, community based programs which provide social support and engagement have been shown to benefit elderly individuals as well as individuals with pathology, but are equally unattainable to this group. Taking the exercise to these individuals via telemedicine or tele-exercise may be an ideal means of delivering this type of intervention.

The long-term goal of this project is to improve outcomes for underserved populations of individuals with Parkinson disease (PD) by providing access to in-home physical activity via a telehealth approach. Approximately one million Americans currently live with a diagnosis of PD and it has been estimated that delaying the progression by 20% would result in a $75,891 savings per individual based on reduced health care costs, income maintenance, increased duration of life and improved quality of life. However, individuals with PD of lower socioeconomic status, people of color and rural dwelling seniors have been critically underserved by clinical and academic programming resulting in poorer health outcomes.

This Study will examine the effects of social engagement during in-home exercise on a small sample of individuals with Parkinson Disease (PD). This pilot investigation will directly measure the effect of social support and engagement on exercise outcomes for rural dwelling individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic "definite PD" based upon established criteria
* vision at or corrected to 20/40 or better
* ability to independently ambulate for at least 10 minutes continuously
* no reported vestibular or neurological disease (stroke or muscle disease) beyond their diagnosed PD
* score of greater than or equal to 78 (no evidence of dementia) on the telephone adaptation of the modified mini-mental state exam
* English Speaking

Exclusion Criteria:

* contraindication for exercise
* history of muscular or orthopedic diagnosis
* inability to participate in the full duration of the study
* currently exercising for 20 or more minutes per week

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen A Pickett, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Dr. Pickett will be responsible for deciding when/to whom to disseminate coded data, and will work with other researchers if necessary to confirm that they have proper IRB approval/etc., as necessary. Required UW-Madison IRB approval would be obtained prior to the release of any data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who started the solo cycling group crossed over to the social cycling group.
Groups:
- Solo Cycling Control Group: Solo Cycling Group: Exercise bike delivered to their home, custom fit to their needs and installed in a safe location. Participants will be provided with exercise recommendations, but will receive only data recording calls every 2-weeks. [will crossover and complete the cycling intervention following the initial 6-months]
Period: Before Crossover to Social Group
Arm/Group | Solo Cycling Control Group | Social Cycling Group
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: After Crossover to Social Group
Arm/Group | Solo Cycling Control Group | Social Cycling Group
Started | 6 | 0
Completed | 6 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One individual assigned to the social cycling group contracted COVID following the baseline assessment and withdrew prior to starting the intervention.
Groups:
- Social Cycling Group Only: Exercise bike delivered to their home, custom fit to their needs and installed in a safe location, sessions will consist of up to 30 minutes of cycling while engaged in social interaction with a research staff member, thus providing a social/community aspect that would not otherwise be present.
  Social Cycling Group: engaged with a research staff member for 30 minutes of cycling
- Total: Total of all reporting groups
Arm/Group | Solo Cycling Control Group | Social Cycling Group Only | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (3.0) | 68.1 (6.9) | 72.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Adherence: Percentage of Sessions Completed
Description: Total number of completed sessions divided by the prescribed number of sessions per study protocol (72)
Time Frame: up to 6 months of active intervention
Population: 12 unique participants, 6 solo cycling group crossed over to social group
Measure: Mean (Full Range); unit: percent sessions completed
Units Other Than Participants: sessions
Arm/Group | Solo Cycling Control Group | Social Cycling Group
Number analyzed (Participants) | 6 | 12
Number analyzed (sessions) | 432 | 864
percent sessions completed | 38.0 [7.0 to 75.0] | 94.6 [88.9 to 98.6]

2. Secondary Outcome: Time Per Session
Description: The number of minutes spent cycling during each session
Time Frame: up to 6 months of active intervention
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Solo Cycling Control Group | Social Cycling Group
Number analyzed (Participants) | 6 | 12
minutes | 16 (11) | 27 (3)

3. Secondary Outcome: Adverse Events
Description: Adverse events that occur during the active intervention period
Time Frame: up to 6 months of active intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Solo Cycling Control Group | Social Cycling Group
Number analyzed (Participants) | 6 | 12
Participants | 0 | 0

4. Other Pre Specified Outcome: Overall Activity Level as Measured by Average Steps Per Day
Description: Participant will wear an activity monitor to collect this data
Time Frame: up to 6 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Canadian Occupational Performance Measure (COPM) Scores
Description: The Canadian Occupational Performance Measure (COPM) will be administered to assess the participant's self-report of performance and satisfaction on a scale of 1 to 10 on self-selected occupational tasks. Performance and satisfaction scores range from 1 (lowest) to 10 (highest) for each identified item. The top three identified occupations will be reported.
Time Frame: baseline, post-test (~6-months)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Fall Frequency
Description: The Fall History Questionnaire is a 6-item survey that asks about Fall rate in the last 2 weeks, last month, last 6 months, the typical cause of a fall, and how the fear of falling may influence daily activities. The hypothesis is that Fall frequency will be improved in the socially engaged cycling group and not with those cycling alone.
Time Frame: baseline, post-test (~6-months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Solo Cycling Control Group | Social Cycling Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 0/6 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT04300023/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT04300023/ICF_001.pdf